CLINICAL TRIAL: NCT04671355
Title: A Phase IV, Open Label, Multicentre, Randomised, 2-way Cross-over Exploratory Clinical Trial Comparing TRIMBOW® pMDI and RELVAR® ELLIPTA® DPI on Lung Stiffness Reduction Assessed Through Area Under the Reactance Curve (AX) in COPD.
Brief Title: TRIMBOW® and RELVAR® on Lung Stiffness Reduction Assessed Through Forced Oscillation Technique in Patients With COPD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Continuing delays due to COVID-19 pandemic
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLI-05993AA1-21; 2019-002744-24 (EudraCT Number)
Record Dates: First submitted 2020-10-28; First posted 2020-12-17 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: COPD
Keywords: Small Airways Disorders and Forced Oscillation Technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone; Formoterol Fumarate; Glycopyrrolate; fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimbow (Experimental): Pressurized metered dose inhaler
  Interventions: Drug: Beclometasone Dipropionate / Formoterol Fumarate / Glycopyrronium 100/6/10 mcg
- Relvar (Active Comparator): Dry powder inhaler
  Interventions: Drug: Fluticasone Furoate / Vilanterol Trifenatate 100/25 mcg

INTERVENTIONS:
Drug: Beclometasone Dipropionate / Formoterol Fumarate / Glycopyrronium 100/6/10 mcg — Pressurized metered dose inhaler
  Arms: Trimbow
Drug: Fluticasone Furoate / Vilanterol Trifenatate 100/25 mcg — Dry powder inhaler
  Arms: Relvar

SUMMARY:
Efficacy of TRIMBOW® pMDI and RELVAR® ELLIPTA® DPI on lung stiffness reduction assessed through area under the reactance curve (AX) using oscillometry in chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
An open label, multicentre, randomised, 2-way cross-over exploratory clinical trial comparing a fixed combination of beclometasone dipropionate plus formoterol fumarate plus glycopyrronium administered via pMDI (TRIMBOW®) and a fixed combination of fluticasone furoate plus vilanterol administered via DPI (RELVAR® ELLIPTA®) on lung stiffness reduction assessed through area under the reactance curve (AX) using forced oscillation technique (FOT) in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent obtained prior to any study related procedures.
2. Male or female patients aged 40 years and above.
3. Patients with established diagnosis of COPD at least 12 months prior to the screening visit (according to GOLD Report, revised 2019). Patients with a diagnosis of Asthma COPD Overlap Syndrome (ACOS) and with a current diagnosis of atopy or allergic rhinitis based on their medical history and investigator judgement will be also eligible for inclusion.
4. Current smokers or ex-smokers, who quit smoking at least 6 months prior to screening visit, with a smoking history of at least 10 pack years [pack-years = (number of cigarettes per day x number of years)/20]. If patients underwent any kind of smoking cessation therapy, it should be finished at least 2 months prior to screening.
5. A post-bronchodilator FEV1 <60 % of the predicted normal value and a post-bronchodilator FEV1/FVC < 0.7 within 30 min after 4 puffs (4 x 100 µg) of salbutamol pMDI.

   If this criterion is not met at screening, the test can be repeated once before randomisation.
6. Patients under double or triple therapy for at least 2 months prior to screening visit in stable doses and regimens with either:

   1. inhaled corticosteroids/long-acting β2-agonist combination (ICS/LABA) (fixed or free), or
   2. inhaled corticosteroids/long-acting muscarinic antagonist free combination (ICS/LAMA), or
   3. Inhaled long-acting β2-agonist / long-acting muscarinic antagonist (LABA/LAMA) (fixed or free), or
   4. fixed or free combination of an inhaled corticosteroid /long-acting β2-agonist/long-acting muscarinic antagonist (ICS/LABA/LAMA)
7. A cooperative attitude and ability to correctly use the study inhalers and spacer.
8. Female patients must be either of non-childbearing potential (WONCBP) defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile) or physiologically capable of becoming pregnant (i.e. women of childbearing potential (WOCBP) fulfilling one of the following criteria:

   1. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up contact or
   2. WOCBP with non-fertile male partners (contraception is not required in this case).For the definition of WONCBP, WOCBP, fertile men, and the list of highly effective birth control methods, refer to Appendix 3 (or section 4.1 of the CTFG guidance).

Any postmenopausal women (physiologic menopause defined as "12 consecutive months of amenorrhea") or women permanently sterilized (e.g. bilateral oophorectomy, hysterectomy or bilateral salpingectomy) may be enrolled in the Study.

Exclusion Criteria:

1. Pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS are willing to use one or more of the highly effective birth control method as reported in Appendix 3 (or section 4.1 of the CTFG guidance).
2. Diagnosis of asthma.
3. Patients requiring use of the following medications:

   i. A course of systemic steroids longer than 3 days for COPD exacerbation in the 4 weeks prior to screening.

   ii. A longer than 7-day course of antibiotics for the treatment of COPD exacerbation in the 4 weeks prior to screening.

   iii. Use of antibiotics for a lower respiratory tract infection (e.g pneumonia) in the 4 weeks prior to screening.
4. COPD exacerbation requiring prescriptions of systemic corticosteroids and/or antibiotics or hospitalization during the run-in period.
5. Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia.
6. Known respiratory disorders other than COPD which may impact the efficacy of the study drug according the investigator's judgment. This can include but is not limited to alfa-1 antitrypsin deficiency, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension and interstitial lung disease.
7. Patients who have clinically severe cardiovascular condition (such as but not limited to unstable ischemic heart disease, NYHA Class III/IV, left ventricular failure, acute myocardial infarction, not controlled arrhythmia etc.), which may impact the efficacy or the safety of the study drug according to the investigator's judgement
8. An abnormal and clinically significant 12-lead ECG which may impact the safety of the patient according to investigator's judgement. Patients whose electrocardiogram (ECG) (12 lead) shows QTcF >450 ms for males or QTcF >470 ms for females at screening or at randomisation visits are not eligible. The QTcF criterion should not be applicable to patients with pacemaker or permanent atrial fibrillation.
9. Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic agents.
10. History of hypersensitivity to anticholinergics, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the trial which may raise contra-indications or impact the efficacy of the study drug according to the investigator's judgement.
11. Clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease which may impact the efficacy or the safety of the study drug according to investigator's judgement.
12. Unstable concurrent disease: e.g. fever, uncontrolled hyperthyroidism, uncontrolled diabetes mellitus or other endocrine disease; significant hepatic impairment; significant renal impairment; uncontrolled gastrointestinal disease (e.g. active peptic ulcer); uncontrolled neurological disease; uncontrolled haematological disease; uncontrolled autoimmune disorders, or other which may impact the efficacy or the safety of the study drug according to investigator's judgment.
13. History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening visit.
14. Participation in another clinical trial where investigational drug was received less than 30 days or 5 half-lives whichever is longer prior to screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-04 (Estimated); Primary Completion 2021-12-22 (Estimated); Study Completion 2022-02-18 (Estimated)

PRIMARY OUTCOMES:
Oscillometry - Reactance (AX) | 4 weeks
  Area under the curve of Reactance (AX) 5-120 minutes post-dose

SECONDARY OUTCOMES:
Oscillometry - Resistance at 5 Hertz (R5) | 4 weeks
  Change from baseline 5-120 minutes post-dose
Spirometry - Forced Expiratory Volume in the first second | 4 weeks
  Change from baseline in pre-dose and post-dose (30, 60 and 120 minutes post-dose)
Health status | 4 weeks
  Change from baseline in COPD Assessment Test (CAT) score
Safety monitoring - incidence of adverse events (AEs) and adverse drug reactions (ADRs) | Overall study period and by Treatments (4 weeks)
  Recording of AEs and ADRs
Oscillometry - Resistance at 19 Hertz (R19) and 20 Hertz (R20) | 4 weeks
  Change from baseline 5-120 minutes post-dose
Oscillometry - Resonance frequency (RF) | 4 weeks
  Change from baseline 5-120 minutes post-dose
Spirometry - Forced Vital Capacity | 4 weeks
  Change from baseline in pre-dose and post-dose (30, 60 and 120 minutes post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lipworth, MD, Study Director — Ninewells Hospital, University of Dundee, Scotland, UK; Catherine Jackson, MD, Principal Investigator — University of Central Lancashire, Burnley, UK

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- See also: EMA Register - EudraCT results section — https://www.clinicaltrialsregister.eu/ctr-search/trial/2019-002744-24/results